CLINICAL TRIAL: NCT05960435
Title: The Effects of Proprioceptive Neuromuscular Facilitation Techniques on Clinical Outcomes in Patients with Proximal Humerus Fractures
Brief Title: Proprioceptive Neuromuscular Facilitation Techniques in Proximal Humerus Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUC35
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PNF group (Experimental): Patients in the PNF group will deliver PNF stretching, active-assistive ROM exercises, PNF scapular patterns mobilization, posterior capsule stretching, and isometric strengthening for 3 weeks. Between 3-6 weeks PNF stretching and scapular mobilization exercises will progress and PNF strengthening and active ROM exercises will add to the program.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation
- Control group (Active Comparator): Patients in the conservative group will deliver shoulder muscle static stretching, active-assistive ROM exercises, scapular mobilization, posterior capsule stretching, and isometric strengthening for 3 weeks. Between 3-6 weeks these exercises will progress and shoulder muscles strengthening via NMES and active ROM exercises will add to the program.
  Interventions: Other: Control Group Exercise

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — PNF, a method used to increase the range of motion of the joint and strengthen the muscles in the newly gained range, is a holistic approach and is based on motor learning principles. PNF stretching involves isometric contraction of the target muscle in addition to static stretching.
  Arms: PNF group
Other: Control Group Exercise — The control group will include static stretching, capsule stretching, progressive ROM exercises and strengthening exercises.
  Arms: Control group

SUMMARY:
The aim of this study is to compare the effect of Proprioceptive Neuromuscular Facilitation (PNF) techniques on functional status, pain, range of motion (ROM), muscle strength, quality of life, and patient satisfaction in people with Proximal Humerus Fracture. There will be two groups, PNF and conservative treatment, and the program will consist of 6 weeks. Patients will randomly be assigned to the conservative treatment group and the PNF group. Patients in the conservative group will deliver shoulder muscle static stretching, active-assistive ROM exercises, scapular mobilization, posterior capsule stretching, and isometric strengthening for 3 weeks. Between 3-6 weeks these exercises will progress and shoulder muscles strengthening via Neuromuscular Electrical Stimulation (NMES) and active ROM exercises will add to the program. Patients in the PNF group will deliver PNF stretching, active-assistive ROM exercises, PNF scapular patterns mobilization, posterior capsule stretching, and isometric strengthening for 3 weeks. Between 3-6 weeks PNF stretching and scapular mobilization exercises will progress and PNF strengthening and active ROM exercises will add to the program.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of Proprioceptive Neuromuscular Facilitation (PNF) techniques on functional status, pain, range of motion (ROM), muscle strength, quality of life, and patient satisfaction in people with Proximal Humerus Fracture. There will be two groups, PNF and conservative treatment, and the program will consist of 6 weeks. Patients will randomly be assigned to the conservative treatment group and the PNF group. Patients in the conservative group will deliver shoulder muscle static stretching, active-assistive ROM exercises, scapular mobilization, posterior capsule stretching, and isometric strengthening for 3 weeks. Between 3-6 weeks these exercises will progress and shoulder muscles strengthening via NMES and active ROM exercises will add to the program. Patients in the PNF group will deliver PNF stretching, active-assistive ROM exercises, PNF scapular patterns mobilization, posterior capsule stretching, and isometric strengthening for 3 weeks. Between 3-6 weeks PNF stretching and scapular mobilization exercises will progress and PNF strengthening and active ROM exercises will add to the program. Measurements will always taken by the blinded therapist who did not deliver the interventions. Our primary outcome measure was the function of the upper limb as assessed by the Turkish version of the Disability of the Arm, Shoulder and Hand (DASH) questionnaire. SF-36 for quality of life andThe Global Rating of Change Scale. (GRC). The outcome assessments will be evaluated at three points in time: at the baseline, after a three-week intervention, and at the end of the treatment (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with humerus proximal fracture and stable information obtained by an orthopedist
* Patients aged ≥ 18 years
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Bad union of tuberculum majus
* Advanced osteoporosis
* Humeral head avascular necrosis
* Presence of severe cardiac disease
* Uncontrollable hypertension
* Presence of neurological and rheumatological disease
* Presence of recurrent infection and open wound incision in the region
* Patients with communication problems
* Patients for whom exercise is not indicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Disability of the Arm, Shoulder and Hand (DASH) questionnaire | 6 weeks
  The DASH is a validated score to assess the physical function and symptoms of people with upper limb disabilities. It contains 30 questions: 6 items about symptoms and 21 items about function. Patients answer the questions using a 5-point, scaling from 0 to 100, with higher scores indicating more disability.

SECONDARY OUTCOMES:
The Constant-Murley (CSM) | 6 weeks
  CSM score evaluates the functional status of the shoulder in patients with shoulder pain. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The maximum total score is 100 points and a high score corresponds to a well-functioning shoulder
Visual Analog Scale (VAS) | 6 weeks
  VAS is used for pain during rest, at night, and during daily activity. In the VAS assessment, the patients are asked to place a vertical mark on a scale where 0 points indicated 'no pain' and 10 points indicated 'worst pain
Range of Motion (ROM) | 6 weeks
  Shoulder flexion, extension, abduction, external and internal rotation will measure with a digital goniometer.
Muscle strength | 6 weeks
  Shoulder flexion, abduction, and scaption in the sitting position, and shoulder internal and external rotation strength will assess by hand-held dynamometer.
The Tampa Scale for Kinesiophobia (TSK) | 6 weeks
  TSK is a 11-item questionnaire used to assess the subjective rating of fear of movement. Each question is scored on a 4-point Likert scale and Total scores range from 11 to 44. High scores indicate an increasing degree of fear of movement.
Short Form-36 (SF-36) | 6 weeks
  The SF-36 questionnaire consists of eight multiple-item subscales that evaluate physical functioning, social functioning and role limitations due to physical problems and role limitations due to emotional problems, mental health, vitality, pain, and general health perception. The total score range from 0 - 100 and higher scores show a better health status.
The Global Rating of Change Scale (GRC) | 6 weeks
  GRC is used for the perception of improvement/deterioration over time. Patients is asked to evaluate their post-treatment status with the 5- point Likert Scale on which -2: much worse, -1: worse, 0: same, +1: better, +2: much better. High scores were positively correlated with satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kus G, Zengin Alpozgen A, Razak Ozdincler A, Gungor F, Altun S. The effectiveness of proprioceptive neuromuscular facilitation techniques versus conventional therapy in patients with proximal humerus fracture: randomized controlled trial. Physiother Theory Pract. 2025 Sep;41(9):1851-1865. doi: 10.1080/09593985.2025.2486418. Epub 2025 Apr 1. PMID 40170293